CLINICAL TRIAL: NCT01189162
Title: High Flow Nasal Cannula Versus Nasal Intermittent Mandatory Ventilation for Respiratory Distress Syndrome: a Randomized, Controlled, Prospective Study
Brief Title: High Flow Nasal Cannula (HFNC) Versus Nasal Intermittent Mandatory Ventilation (NIMV)for Respiratory Distress Syndrome (RDS): a Randomized, Controlled, Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31/09
Record Dates: First submitted 2010-08-23; First posted 2010-08-26 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Distress Syndrome
Keywords: Primary treatment of RDS and treatment of RDS post extubation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIMV- nasal respiratory support (Experimental): Infants with RDS will be treateg with nasal intermittent mandatory ventilation
  Interventions: Device: NIMV with SLE ventilator vs HFNC via Vapotherm
- HFNC- nasal respiratory support with HFNC (Experimental): Infants with RDS will be treated with nasal respiratory support with high flow nasal canulla
  Interventions: Device: NIMV with SLE ventilator vs HFNC via Vapotherm

INTERVENTIONS:
Device: NIMV with SLE ventilator vs HFNC via Vapotherm — Nasal respiratory support for RDS
  Other Names: NIMV with SLE ventilator vs. HFNC via Vapotherm

SUMMARY:
The investigators hypothesize that while the extremely low birthweight (ELBW) infants (<1000 g) may need NIMV for the treatment of RDS, larger infants or the smaller ones post extubation may enjoy the comfort benefits associated with HFNC while getting coparable respiratory support to NIMV.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age between 24 to 34 and 6/7 weeks assessed by the obstetrical team from dating of last menstural period or ultrasound and weight >1000 g for the initial treatment of RDS or <35 weeks post extubation or for apnea of prematurity
2. Infants with RDS who will need NRS as initial therapy or after extubation and for apnea of prematurity, 3. written informed consent.

Exclusion Criteria:

1. Significant morbidity apart from RDS including: cardiac disease (not including patent ductus arteriosus [PDA]), congenital malformation, or if they had cardiovascular or respiratory instability because of sepsis, anemia or severe intraventricular hemorrhage (IVH),
2. Parents refuse consent.
3. Unavailability of suitable ventilator.

Min Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The percent of infants who will fail NRS and need endotracheal ventilation or will be switched to another mode of NRS. | 1 year

SECONDARY OUTCOMES:
Clinical features on both methods | 1 year
  Blood pressure, heart rate, respiratory rate, pulse oximetry saturation, and respiratory status prior to mechanical ventilation if needed according to arterial blood gas (PaO2, PCO2, pH), and "time to stop nasal support"
% of infants with neonatal morbidities on both methods | 1 year
  Incidence of intraventricular hemorrhage (IVH), duration of mechanical ventilation, incidence of BPD (oxygen at 36 weeks post conceptional age to keep saturation>92%), time until full feeds, and length of stay.
% of infants with possible side effects on both methods | 1 year
  Nasal trauma due to NRS, rate of air leak (pneumothorax), gastrointestinal perforation, irritability and discomfort assessed by a validated score

CONTACTS AND LOCATIONS:
Overall Officials: Amir Kugelman, MD, Principal Investigator — Bnai Zion Medical Cente
Locations (1):
- Bnai Zion Medical Center, Neonatal department, Haifa, Israel

REFERENCES:
- [Background] Kugelman A, Feferkorn I, Riskin A, Chistyakov I, Kaufman B, Bader D. Nasal intermittent mandatory ventilation versus nasal continuous positive airway pressure for respiratory distress syndrome: a randomized, controlled, prospective study. J Pediatr. 2007 May;150(5):521-6, 526.e1. doi: 10.1016/j.jpeds.2007.01.032. PMID 17452229
- [Derived] Kugelman A, Riskin A, Said W, Shoris I, Mor F, Bader D. A randomized pilot study comparing heated humidified high-flow nasal cannulae with NIPPV for RDS. Pediatr Pulmonol. 2015 Jun;50(6):576-83. doi: 10.1002/ppul.23022. Epub 2014 Mar 12. PMID 24619945